CLINICAL TRIAL: NCT00529607
Title: New Imaging and Diagnostic Techniques for the Assessment of Reperfusion Injury in Myocardial Infarction.
Brief Title: Diagnostics for the Reperfusion Injury Following MI
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: RWTH Aachen University, Medical Clinic I and IZKF Biomat
Other Study IDs: IZKF BIOMAT Aachen TVB 119
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Reperfusion Injury
Keywords: myocardial infarction, reperfusion injury, echocardiography, magnetic resonance imaging, inflammation, nitric oxide
MeSH Terms: conditions — Reperfusion Injury; Myocardial Infarction; Inflammation | interventions — perflutren; contrast agent BR1; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomarkers for Infarction and Inflammation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: - patients with acute ST elevation myocardial infarction and consecutive percutaneous coronary intervention of the infarct-related artery
  Interventions: Drug: contrast echocardiography; Procedure: 2D and 3D echocardiography; Procedure: cardiac MRI; Procedure: blood sampling
- 2: - 30 patients with stable CAD (control group 1)
  Interventions: Procedure: blood sampling
- 3: - 30 healthy volunteers regarding cardiovascular diseases (control group 2)
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Drug: contrast echocardiography — directly after PCI, at 24 h after PCI, before discharge and at 6 months
  Other Names: with luminity or sonovue
  Groups: 1
Procedure: 2D and 3D echocardiography — directly after PCI, at 24 h after PCI, before discharge and at 6 months
  Groups: 1
Procedure: cardiac MRI — before discharge and after 6 months
  Groups: 1
Procedure: blood sampling — routine lab work plus infarction and inflammation biomarkers
  1: before PCI, after PCI, at 34 hours, at discharge, at 6 months 2 and 3: one blood sample in total before PCI in 2 and at any time in 3

SUMMARY:
The primary purpose of this study is to correlate new cardiac imaging modalities (2D, 3D echocardiography, contrast echocardiography, strain analysis and cardiac MRI) to biochemical parameters as the L-arginine-nitric oxide pathway and inflammatory cascades to characterize the reperfusion injury following myocardial infarction and thus providing a basis for further diagnostic and therapeutic approaches.

DETAILED DESCRIPTION:
By reperfusion of ischemic myocardium further tissue damage occurs (ischemia / reperfusion injury). Various contributing mechanisms have been discussed in experimental studies, e.g. disturbances in coronary microcirculation and consecutive induction of inflammatory cascades involving formation of reactive oxygen species. The ischemia / reperfusion injury causes diastolic and regional as well as global systolic dysfunction. The time course of the reperfusion injury within the first hours after reperfusion and its effects on the global geometry of the left ventricle have not been investigated so far. In the present study a comprehensive morphological and functional characterisation of the ischemia / reperfusion injury in the acute phase is performed. New cardiac imaging modalities (2D, 3D echocardiography, contrast echocardiography, strain analysis and cardiac MRI)and biochemical parameters including the L-arginine-nitric oxide pathway and inflammatory cascades are applied. Hereby morphological and biochemical markers for the functional recovery of myocardial function should be identified.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute ST elevation myocardial infarction and consecutive percutaneous coronary intervention of the infarct-related artery (first myocardial infarction and recurrent myocardial infarction, as long as infarct-related artery is occluded for the first time)
* written informed consent

or 30 patients with stable CAD (control group 1) or 30 healthy volunteers regarding cardiovascular diseases (control group 2)

Exclusion Criteria:

* minors
* incompetent persons
* pregnant and lactating
* moderate to severe renal insufficiency defined by an GFR < 60 ml/kg/m2
* missing written consent
* other reasons complicating a clinical reevaluation and/or coronary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * patients with acute ST elevation myocardial infarction and consecutive percutaneous coronary intervention of the infarct-related artery (first myocardial infarction and recurrent myocardial infarction, as long as infarct-related artery is occluded for the first time)
  * written informed consent
  or 30 patients with stable CAD (control group 1) or 30 healthy volunteers regarding cardiovascular diseases (control group 2)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Lepper, Principal Investigator — Department of Medicine, Division of Cardiology, Pulmonary Diseases and Vascular Medicine at the University Hospital, RWTH Aachen
Locations (1):
- Department of Medicine, Division of Cardiology, Pulmonary Diseases and Vascular Medicine at the University Hospital, RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Kehmeier ES, Lepper W, Kropp M, Heiss C, Hendgen-Cotta U, Balzer J, Neizel M, Meyer C, Merx MW, Verde PE, Ohmann C, Heusch G, Kelm M, Rassaf T. TNF-alpha, myocardial perfusion and function in patients with ST-segment elevation myocardial infarction and primary percutaneous coronary intervention. Clin Res Cardiol. 2012 Oct;101(10):815-27. doi: 10.1007/s00392-012-0465-x. Epub 2012 May 6. PMID 22562290